CLINICAL TRIAL: NCT02841423
Title: Postoperative Cognitive Dysfunction After Intravenous Anesthesia or Closed-loop Coadministration of Propofol and Remifentanil Guided by Bispectral Index for Noncardiac Surgery : a Randomized Monocenter Study
Brief Title: Postoperative Cognitive Dysfunction After Propofol Anesthesia for Noncardiac Surgery
Acronym: POCD ELA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: API/2013/44
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Patients ASA I, II, III
Keywords: physical status I-III;; age > 55 yr); undergoing surgery (duration, > 1 h)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INTRAVENOUS ANESTHESIA (Experimental): neuropsychological test battery
  Interventions: Procedure: neuropsychological test battery
- CLOSED LOOP ANESTHESIA (Experimental): neuropsychological test battery
  Interventions: Procedure: neuropsychological test battery

INTERVENTIONS:
Procedure: neuropsychological test battery

SUMMARY:
Background: Postoperative cognitive dysfunction (POCD) in elderly patients after noncardiac surgery is a common problem.

Therefore,this study was designed to assess POCD after closed-loop coadministration of propofol and remifentanil guided by bispectral index in comparison to intravenous anesthesia in elderly patients undergoing major noncardiac surgery. Methods: After approval of the local ethical committee was obtained, 204 patients (American Society of Anesthesiologists physical status I-III; age, > 55 yr) undergoing surgery (duration, > 1 h) were enrolled into this pospective randomized monocenter study. Patients received anesthesia 3 days after using a neuropsychological test battery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-III;
* undergoing surgery (duration, > 1 h)

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-08 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
the incidence of early POCD in elderly patients (aged 55 yrs or older) | 3 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: E SAMAIN, PR, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- Chu Besancon, Besançon, France

REFERENCES:
- [Derived] Besch G, Vettoretti L, Claveau M, Boichut N, Mahr N, Bouhake Y, Liu N, Chazot T, Samain E, Pili-Floury S. Early post-operative cognitive dysfunction after closed-loop versus manual target controlled-infusion of propofol and remifentanil in patients undergoing elective major non-cardiac surgery: Protocol of the randomized controlled single-blind POCD-ELA trial. Medicine (Baltimore). 2018 Oct;97(40):e12558. doi: 10.1097/MD.0000000000012558. PMID 30290615